CLINICAL TRIAL: NCT02424526
Title: Intensive Home-based Treadmill Training and Walking Attainment in Young Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Sacramento (Other)
Collaborators: Seattle Children's Hospital (Other); University of Puget Sound (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Katrin Mattern-Baxter, PT, DPT, PCS, California State University, Sacramento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-14-156
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; treadmill training; walking
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high-intensity group (Active Comparator): Children will engage in home-based treadmill training 5 days/week, twice daily for 10-20 min for 6 weeks
  Interventions: Other: home-based treadmill training; Device: Treadmill
- low-intensity group (Active Comparator): Children will engage in home-based treadmill training 2 days/week, once daily for 10-20 minutes for 6 weeks
  Interventions: Other: home-based treadmill training; Device: Treadmill

INTERVENTIONS:
Other: home-based treadmill training — the child will walk on a pediatric treadmill with the help of the parent/caregiver and with weekly supervision of a physical therapist
Device: Treadmill

SUMMARY:
This study is designed to find the optimal dosage of home-based treadmill training needed to accelerate walking onset and to examine the long-term effects on the child's walking activity.

DETAILED DESCRIPTION:
The purpose of this study is to determine optimal parameters for dosing home-based treadmill training by comparing high-intensity (5 days/week, twice daily for 10-20 min for 6 weeks) to low-intensity (2 days/week, once daily for 10-20 minutes for 6 weeks) treadmill training; and to compare the effects of high- versus low-intensity treadmill training on walking attainment and overall walking activity in young children with cerebral palsy.

Hypotheses

* A more intensive protocol of treadmill training will increase walking onset in young children with CP.
* A more intensive protocol of treadmill training will increase overall walking activity in young children with CP.

Specific Aims

* To determine optimal parameters for dosing home-based treadmill training by comparing high-intensity to low-intensity home-based treadmill training.
* To compare the effects of high- versus low-intensity treadmill training on walking onset and overall walking activity.

Study design •Prospective randomized controlled trial

Study population

•Two groups of 12 children with CP under the age of 3 years and are not walking yet will receive either home-based high-intensity treadmill training or low-intensity treadmill training. The children will be assessed before, immediately after, at 1-month and at 4-months following the intervention via standardized outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Signs of walking readiness as demonstrated by the ability to sit for 30 seconds when placed and to take 5 to 7 steps when supported at the trunk or arms.
* Because young children often are not formally diagnosed with CP until 2 years of age, we will include children

  * who show bilateral impairment (i.e. diplegia and quadriplegia, but not hemiplegia)
  * who demonstrate upper motor neuron signs (i.e. spasticity and/or hyperreflexia)
  * who have been identified as high-risk for a motor disability by a physician

Exclusion Criteria:

* a history of uncontrolled seizures
* a diagnosis of a genetic disorder
* cardiac or orthopedic contraindications for standing and walking
* orthopedic surgery in the past 6 months
* use of spasticity-reducing medication or Botox injections in the past 6 months

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Earwicker, BA,MA, Study Director — California State University, Sacramento
Locations (2):
- United States (2):
  - Seattle Children's Research Institute, Seattle, Washington
  - University of the Puget Sound, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattern-Baxter K, Looper J, Zhou C, Bjornson K. Low-Intensity vs High-Intensity Home-Based Treadmill Training and Walking Attainment in Young Children With Spastic Diplegic Cerebral Palsy. Arch Phys Med Rehabil. 2020 Feb;101(2):204-212. doi: 10.1016/j.apmr.2019.09.015. Epub 2019 Nov 1. PMID 31678223

RESULTS

PARTICIPANT FLOW:
Groups:
- High-intensity Group: Children will engage in home-based treadmill training 5 days/week, twice daily for 10-20 min for 6 weeks
  home-based treadmill training: the child will walk on a pediatric treadmill with the help of the parent/caregiver and with weekly supervision of a physical therapist
  Treadmill
- Low-intensity Group: Children will engage in home-based treadmill training 2 days/week, once daily for 10-20 minutes for 6 weeks
  home-based treadmill training: the child will walk on a pediatric treadmill with the help of the parent/caregiver and with weekly supervision of a physical therapist
  Treadmill
Period: Overall Study
Arm/Group | High-intensity Group | Low-intensity Group
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data from one participant could not be analyzed after post-test due to Botox injections.
Groups:
- High-intensity Group: High-intensity engaged in treadmill training 10x/week for 6 weeks
- Low-intensity Group: Low-intensity engaged in treadmill training 2x/week for 6 weeks
- Total: Total of all reporting groups
Arm/Group | High-intensity Group | Low-intensity Group | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 10 | 19
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 2 | 2 | 4
  Asian | 1 | 1 | 2
  Hispanic | 2 | 1 | 3
  White | 2 | 5 | 7
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Gross Motor Function Measure Dimension E
Description: The Gross Motor Function Measure is a criterion-referenced test of gross motor function for children with cerebral palsy ages 5 months to 15 years. It contains 5 Dimensions (A-E). Dimension E is related to the child's gross motor skills related to walking, running and jumping and is assessed by observation. Dimension E contains 24 gross motor skills. Each of these motor skills is rated either 0 (does not initiate), 1(initiates), 2 (partially completes), 3 (completes) or NT( not tested). The total possible Dimension E score is 72 with a range of 0-72. Scores can be converted into a percent score by dividing the child's achieved points by the number of possible points. Higher scores and a higher percentage indicate better performance in walking, running and jumping. Change from baseline in total points, not in percentage, is reported.
Time Frame: assessed at 6 weeks, 1 month, 4 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
score on a scale
  6 weeks | 15.6 (5.9) | 12.7 (9.7)
  1 month | 18.7 (7.5) | 17.1 (8.8)
  4 months | 16.2 (5.9) | 14.1 (7.7)

2. Primary Outcome: Walking Activity Measured by StepWatch
Description: StepWatch data records the child's walking activity in minutes/day. It is collected via an accelerometer attached to the distal leg and worn at all waking hours except during sleep and bath time.Higher numbers of active minutes indicate higher level of activity. Changes from baseline are reported.
Time Frame: StepWatch data was collected for all awake daytime hours over a 7 day period at study onset before treadmill training commences and at 6 weeks, 1 month, 4 months.
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- High-intensity Group: treadmill training 10x/week
- Low-intensity Group: treadmill training 2x/week
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
minutes
  6 weeks | 39.43 [-60.76 to 139.6] | 25.09 [-5.02 to 55.20]
  1 month | 83.33 [-20.80 to 187.46] | 18.01 [-12.10 to 48.12]
  4 months | 132.00 [27.86 to 236.14] | 41.19 [7.17 to 75.21]

3. Primary Outcome: Gross Motor Function Measure Dimension D
Description: The Gross Motor Function Measure is a criterion-referenced test of gross motor function for children with cerebral palsy ages 5 months to 15 years. It contains 5 Dimensions (A-E).Dimension D is a test of gross motor function related to standing ability. The child's gross motor skills related to standing are assessed by observation. The test contains 13 gross motor skills. Each of these motor skills is rated either 0 (does not initiate), 1(initiates), 2 (partially completes), 3 (completes) or NT( not tested). The total possible Dimension D score is 39 with a range of 0-39. Scores can be converted into a percent score by dividing the child's achieved points by the number of possible points. Higher scores and a higher percentage indicate better performance in standing. Change from baseline in total points, not in percentage, is reported.
Time Frame: assessed at 6 weeks, 1 month, 4 months from baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
score on a scale
  6 weeks | 5.11 [1.05 to 9.17] | 5.30 [2.37 to 8.23]
  1 month | 8.22 [4.16 to 12.28] | 8.72 [5.67 to 11.76]
  4 months | 12.67 [8.60 to 16.73] | 12.94 [9.89 to 15.99]

4. Secondary Outcome: Pediatric Evaluation of Disability Index-Mobility Subscale
Description: The Pediatric Evaluation of Disability Index is a valid and reliable tool that provides an assessment of a child's functional status and performance via observation and parent report.The Mobility Subscale examines the child's functional skills related to movement. There are a total of 13 motor categories on the Mobility Subscale, with 5 possible motor skills in each category, for a total of 65 distinct motor skills. Skills are marked as 0 (not observed) or 1 (observed) and added.There are a total of 65 possible points with a range of 0-65 points on the Mobility Subscale. Higher scores indicate greater function.Scores are reported as changes from baseline.
Time Frame: pre-intervention, at 6 weeks, at 1-month and at 4-months following the intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
score on a scale
  6 weeks | 3.80 [1.41 to 6.1] | 5.44 [1.81 to 9.0]
  1 month | 6.89 [3.26 to 10.00] | 7.51 [5.03 to 10.00]
  4 months | 11.63 [9.14 to 14.11] | 14.00 [10.37 to 17.63]

5. Secondary Outcome: Timed 10-meter Walk Test
Description: The child's walking speed is recorded over 10 meters if the child is able to walk with or without an assistive device. The speed is timed and reported in seconds. Fewer seconds indicate a faster walking speed. Time in seconds is reported as change from baseline.
Time Frame: assessed at 6 weeks, at 1-month and at 4-months following the intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
seconds
  6 weeks | -24.86 [-44.12 to -5.60] | -36.23 [-62.66 to -9.81]
  1 month | -28.16 [-47.42 to -8.90] | -49.65 [-77.01 to -22.12]
  4 months | -46.99 [-66.25 to -27.73] | -38.80 [-66.25 to -11.36]

6. Secondary Outcome: Peabody Developmental Motor Scales-2 -Locomotion Subscale
Description: Peabody Developmental Motor Scales-2 is a norm-referenced standardized test of gross and fine motor performance for children from birth through age 5.The Locomotion Subscale examines the ability of the child to move through space. It contains a total of 89 motor skills. The child is rated on each skill on a scale of 0 (unable), 1 (partial) or 2 (complete) and the scores are added for a total possible raw score of 178 and a range of 0-178. Higher raw scores indicate a better outcome.The raw scores can be converted to standard scores, age equivalents and percentiles Raw scores of the Locomotion subscale are reported based on changes from baseline.
Time Frame: assessed at 6 weeks, at 1-month and at 4-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
score on a scale
  6 weeks | 5.67 [0.88 to 10.46] | 6.70 [3.18 to 10.22]
  1 month | 8.33 [3.55 to 13.12] | 9.21 [5.55 to 12.88]
  4 months | 14.11 [9.32 to 18.90] | 13.99 [10.33 to 17.65]

7. Secondary Outcome: 1-minute Walk Test
Description: The child's walking distance is measured in meters over 1 minute at their self-selected walking speed if the child is able to walk with or without an assistive device.The walking distance is reported in meters. More meters indicate more distance covered. Values are reported in meters as changes from baseline.
Time Frame: assessed at 6 weeks, 1 month, 4 months
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | High-intensity Group | Low-intensity Group
Number analyzed (Participants) | 9 | 10
meters
  6 weeks | 8.28 [3.49 to 13.09] | 7.87 [1.78 to 13.96]
  1 month | 12.38 [7.58 to 17.18] | 9.48 [3.15 to 15.80]
  4 months | 15.37 [10.57 to 20.17] | 16.15 [9.83 to 22.47]

ADVERSE EVENTS:
Time Frame: pre-intervention, at 6 weeks, at 1-month and at 4-months following the intervention.
Description: fatigue, injury, fall, parent-reported or observed
Arm/Group | High-intensity Group | Low-intensity Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
Power analysis was carried out to determine the sample size, however the population for the basis of power analysis was not as homogeneous as the subjects in this study. Not all outcome measures could be blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02424526/Prot_SAP_000.pdf